CLINICAL TRIAL: NCT01788826
Title: Randomized Clinical Trial to Evaluate the Use of a Prophylactic Polypropylene Mesh To Reduce the Incidence of Ventral Hernias in Colorectal Surgery
Brief Title: Prophylactic Mesh to Reduce The Incidence of Ventral Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henares University Hospital (Other)
Responsible Party: Principal Investigator, Miguel A ngel Garci-a Urena, Professor, Henares University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HH01
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2013-02

CONDITIONS: Ventral Hernia
Keywords: Ventral hernia; surgical meshes; polypropylenes
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prophylactic Mesh (Experimental): Use of a prefascial polypropylene mesh when closing midline laparotomy
  Interventions: Procedure: Prophylactic mesh
- No prophylactic mesh closure (Experimental): In this arm the laparotomy of the patients are closed with a running absorbable suture without a mesh
  Interventions: Procedure: No prophylactic mesh closure

INTERVENTIONS:
Procedure: Prophylactic mesh — Closure of midline laparotomy using a prophylactic mesh. The midline is closed with a running absorbable monofilament suture with a suture/wound length ratio 4:1. The material is a monofilament uncoated suture made of poly-4hiydroxybutirate (Monomax, B.Braun) USP 1. Then, a prefascial large-pore low-weight 5 cm wide polypropylene mesh (Optilene Mesh Elastic, B.Braun) is fixed covering the midline closure. The mesh is fixed in the prefascial plane with absorbable monofilament interrupted sutures, USP 2/0.
  Arms: Prophylactic Mesh
Procedure: No prophylactic mesh closure — Closure of midline laparotomy without mesh. The laparotomy is closed with a running absorbable monofilament suture with a suture/wound length ratio 4:1. The material is a monofilament uncoated suture made of poly-4hiydroxybutirate (Monomax, B.Braun) USP 1.
  Arms: No prophylactic mesh closure

SUMMARY:
The incidence of ventral hernias has remained inappropriately high. Any innovation in order to reduce this incidence would be simply cost-effective. Although there is still some concern about the use of mesh in clean-contaminated or contaminated surgery, based in our experimental studies, we plan to use a mesh in the primary closure of abdominal incision to prevent incisional hernias.

The investigators propose a clinical trial to assess a model to prevent the incisional hernia after laparotomy to treat colorectal carcinoma is scheduled. A simple randomization is scheduled: in the intervention group a prefascial large-pore low-weight 5 cm wide polypropylene mesh is fixed covering the midline closure; in the control group a conventional closure with a running suture of long-term absorbable material with a suture/wound length ratio 4:1. The sample size was calculated with an estimated incidence of ventral hernia of 25% in the control group and 10% in the intervention group, 0,05 alfa and a 0,15 beta error. The main goal is the appearance of a ventral hernia after 24 months of follow-up. Other outcomes are wound complications and morbidity. Exclusion criteria are adult patients with a previous ventral hernia, estimated survival of less than 6 months or hemodynamic instability during surgery.

The diagnosis of ventral hernia will be assessed by clinical exploration on 3,6,12,18 and 24 months and abdominal CT controls at 6,12, and 24 months. The study will be statistically evaluated with SPSS 18.0.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years old.
* Patients operated with elective or emergency midline laparotomy with the diagnosis of colorectal cancer.
* Written informed consent or oral consent with the present of two witnesses who do not participate as investigators in the trial

Exclusion Criteria:

* Dissemination of oncologic disease: all stage IV tumors with estimated survival less than 3 months.
* Simultaneous participation in another trial with interference of intervention and outcome.
* Withdrawn or missing written consent.
* Mental condition rendering the subject incapable of understanding the nature, scope and consequences of the trial.
* Previous ventral hernia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Compare the incidence of ventral hernia between the 2 groups | 24 months
  Compare the incidence of ventral hernias at the end of the second year follow-up in patients operated for laparotomy using two different methods of abdominal wall closure: one with mesh reinforcement and another one with no mesh reinforcement

SECONDARY OUTCOMES:
Incidence of superficial surgical site infection | 30 days
  Compare the incidence of superficial surgical site infection between the 2 groups
Incidence of deep surgical site infection | 30 days
  Compare the incidence of deep surgical site infection between the 2 groups
Seroma | 30 days
  Incidence of postoperative seroma
Postoperative complications | 30 days
  Register of postoperative complications, including pulmonary, fistula and postoperative ileum

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Ángel García-Ureña, Professor, Principal Investigator — Henares University Hospital
Locations (1):
- Henares University Hospital, Coslada, Madrid, Spain

REFERENCES:
- [Background] Strzelczyk JM, Szymanski D, Nowicki ME, Wilczynski W, Gaszynski T, Czupryniak L. Randomized clinical trial of postoperative hernia prophylaxis in open bariatric surgery. Br J Surg. 2006 Nov;93(11):1347-50. doi: 10.1002/bjs.5512. PMID 17006977
- [Background] Stringer RA, Salameh JR. Mesh herniorrhaphy during elective colorectal surgery. Hernia. 2005 Mar;9(1):26-8. doi: 10.1007/s10029-004-0274-x. Epub 2004 Sep 10. PMID 15365881
- [Background] Gutierrez de la Pena C, Medina Achirica C, Dominguez-Adame E, Medina Diez J. Primary closure of laparotomies with high risk of incisional hernia using prosthetic material: analysis of usefulness. Hernia. 2003 Sep;7(3):134-6. doi: 10.1007/s10029-003-0124-2. Epub 2003 Apr 3. PMID 12687426
- [Background] O'Hare JL, Ward J, Earnshaw JJ. Late results of mesh wound closure after elective open aortic aneurysm repair. Eur J Vasc Endovasc Surg. 2007 Apr;33(4):412-3. doi: 10.1016/j.ejvs.2006.11.015. Epub 2006 Dec 11. PMID 17164090
- [Background] Bellon JM, Lopez-Hervas P, Rodriguez M, Garcia-Honduvilla N, Pascual G, Bujan J. Midline abdominal wall closure: a new prophylactic mesh concept. J Am Coll Surg. 2006 Oct;203(4):490-7. doi: 10.1016/j.jamcollsurg.2006.06.023. Epub 2006 Aug 23. PMID 17000392
- [Background] Israelsson LA, Millbourn D. Closing midline abdominal incisions. Langenbecks Arch Surg. 2012 Dec;397(8):1201-7. doi: 10.1007/s00423-012-1019-4. Epub 2012 Nov 11. PMID 23143146
- [Background] Diaz-Godoy A, Garcia-Urena MA, Lopez-Monclus J, Vega Ruiz V, Melero Montes D, Erquinigo Agurto N. Searching for the best polypropylene mesh to be used in bowel contamination. Hernia. 2011 Apr;15(2):173-9. doi: 10.1007/s10029-010-0762-0. Epub 2010 Dec 9. PMID 21152940